CLINICAL TRIAL: NCT00989846
Title: Feasibility Study on Establishing Biomarkers in Lung Diseases
Brief Title: Biomarker in Lung Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Dr. Michael Kreuter, Thoraxklinik Heidelberg
Other Study IDs: MK02
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Lung Diseases
Keywords: biomarker; lung disease
MeSH Terms: conditions — Lung Diseases | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum (blood)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lung disease: patients with various chronic or acute lung diseases
  Interventions: Other: biomarker

INTERVENTIONS:
Other: biomarker — measuring serum-biomarkers

SUMMARY:
Disease related biomarkers have been established decades ago, e.g. blood glucose for diabetes diagnosis and management. Their discovery has grown dramatically during the past decade and they have the potential to lead the physician in diagnosis -especially differential diagnosis - and therapy.

However, a specific serum-biomarker in lung diseases has not been established. Aim of the current study is to to measure lung specific proteins in the serum in patients with various lung diseases and to correlate those with disease severity, lung function and other laboratory results

ELIGIBILITY:
Inclusion Criteria:

* age >= 18
* acute or chronic lung disease

Exclusion Criteria:

* HIV
* lactation or gestation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute or chronic lung diseases
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-03 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Serum biomarker expression | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kreuter, MD, Principal Investigator — Thoraxklinik Heidelberg, Germany; Felix JF Herth, MD, Study Director — Thoraxklinik Heidelberg Germany
Locations (1):
- Thoraxklinik Heidelberg, Dept. of Pneumology and Respiratory Critical care, Heidelberg, Germany

REFERENCES:
- [Background] Tzouvelekis A, Pneumatikos I, Bouros D. Serum biomarkers in acute respiratory distress syndrome an ailing prognosticator. Respir Res. 2005 Jun 22;6(1):62. doi: 10.1186/1465-9921-6-62. PMID 15972108
- [Background] Tzouvelekis A, Kouliatsis G, Anevlavis S, Bouros D. Serum biomarkers in interstitial lung diseases. Respir Res. 2005 Jul 21;6(1):78. doi: 10.1186/1465-9921-6-78. PMID 16042760